CLINICAL TRIAL: NCT00426556
Title: A Phase Ib/II Study Investigating the Combination of Everolimus With Trastuzumab and Paclitaxel in Patients With HER2-overexpressing Metastatic Breast Cancer
Brief Title: Efficacy and Safety of Everolimus in Combination Therapy, in Patients With HER2-overexpressing Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001J2101; 2006-001596-37 (EudraCT Number)
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Cancer of the breast; Human mammary carcinoma; HER-2; Metastatic; everolimus; trastuzumab; paclitaxel
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Everolimus; Trastuzumab; Paclitaxel

ARMS (4):
- Phase I - RAD001 5mg + PT, daily (Experimental): Daily dosing schedule of EPT = Paclitaxel & Trastuzumab verolimus 5mg plus Paclitaxel plus Trastuzumab.
  Interventions: Drug: Everolimus; Drug: Trastuzumab; Drug: Paclitaxel
- Phase I - RAD001 10mg + PT, daily (Experimental): Daily dosing schedule of Everolimus 10mg plus Paclitaxel plus Trastuzumab. PT = Paclitaxel & Trastuzumab
  Interventions: Drug: Everolimus; Drug: Trastuzumab; Drug: Paclitaxel
- Phase I - RAD001 30mg + PT, weekly (Experimental): Weekly dosing schedule of Everolimus 30mg plus Paclitaxel plus Trastuzumab. PT = Paclitaxel & Trastuzumab.
  Interventions: Drug: Everolimus; Drug: Trastuzumab; Drug: Paclitaxel
- Phase II - RAD001 10mg + PT, daily (Experimental): Daily dosing schedule of Everolimus 10mg plus Paclitaxel plus Trastuzumab. PT = Paclitaxel & Trastuzumab
  Interventions: Drug: Everolimus; Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Everolimus — Everolimus (RAD001) was supplied as tablets in 3 different dosage strengths, 2.5, 5, and 10 mg. The drug was packaged in blisters containing 10 tablets per blister. Blisters and packaging labels were compliant with local regulations and were printed in local language.
  Other Names: RAD001
Drug: Trastuzumab — Commercially-available trastuzumab was used in this study. A 4 mg/kg loading dose was administered, intra-venous (IV), over 90 minutes on Day 1 (if patient was not already receiving trastuzumab); this was followed by weekly trastuzumab 2 mg/kg IV administered over 30 minutes. For patients who continued to receive trastuzumab and everolimus after completion/discontinuation of chemotherapy in the core treatment phase, trastuzumab may have been administered once every 3 weeks at a dose of 6 mg/kg. PT = Paclitaxel & Trastuzumab
Drug: Paclitaxel — Commercially-available paclitaxel was used in this study. Paclitaxel infusion was administered on Days 1, 8, and 15 of each 28-day cycle, after administration of trastuzumab. Paclitaxel (80 mg/m2) was administered as a 60-minute continuous IV infusion after standard premedication. Patients received paclitaxel for 6 cycles. At the investigator's discretion, treatment with paclitaxel could continue beyond 6 cycles.

SUMMARY:
Phase I: will look at different dose levels and regimens of everolimus combined with weekly trastuzumab and paclitaxel therapy in patients with HER-2 overexpressing metastatic breast cancer.

Phase II: will assess the efficacy and safety of the 10mg daily dose of everolimus combined with weekly trastuzumab and paclitaxel therapy in patients with HER-2 overexpressing metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients ≥ 18 years old with WHO performance status ≤ 1
* HER-2 over-expressing metastatic breast cancer cells confirmed by histology
* Progressive disease on prior trastuzumab alone/or in combination with other anticancer agents, or relapsed any time after completion of this therapy (phase l)
* Patient resistance to trastuzumab and taxanes (Phase ll)
* Measurable disease according to RECIST (Phase ll)
* Patients neurologically stable with adequate bone marrow, liver and renal function

Exclusion Criteria:

* Patients receiving endocrine therapy for breast cancer ≤ 2 weeks prior to study treatment start
* Patients currently receiving chemotherapy, immunotherapy or radiotherapy or who have received these ≤ 4 weeks prior to study treatment start or patients who have received lapatinib ≤ 2 weeks prior to study treatment start
* Patients who have previously received mTOR inhibitors

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- United States (11):
  - Wilshire Oncology Medical Group La Verne, *see Various Departments*, California
  - Compassionate Cancer Care Medical Group Dept.ofCCCMG, Fountain Valley, California
  - Loma Linda University Dept.ofLomaLindaCancerCent(3), Loma Linda, California
  - University of California at Los Angeles Dept.of UCLA Dept.ofMed., Los Angeles, California
  - Florida Cancer Research Institute, Davie, Florida
  - Emory University School of Medicine/Winship Cancer Institute Dept. of Hematology (2), Atlanta, Georgia
  - North Shore University Health System, Evanston, Illinois
  - Peninsula Regional Medical Center Deptof Oncology and Hematology, Salisbury, Maryland
  - Washington University School Of Medicine-Siteman Cancer Ctr StudyCoordinator:CRAD001J2101, St Louis, Missouri
  - Cancer Centers of the Carolinas CC of C -Eastside, Greenville, South Carolina
  - Sammons Cancer Center - Texas Oncology, Dallas, Texas
- Belgium (3):
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Turnhout
- France (4):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Maastricht, Netherlands
- Novartis Investigative Site, Lleida, Catalonia, Spain

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=712

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on the results of the Phase I portion of this study, in addition to all available information on daily and weekly everolimus regimen in breast cancer and other tumors, all patients in the Phase II portion of the study were allocated to one arm to receive the recommended everolimus dose of 10 mg daily in combination with PT.
Groups:
- Phase I - RAD001 5mg + PT, Daily: Daily dosing schedule of Everolimus 5mg plus Paclitaxel plus Trastuzumab. PT = Paclitaxel & Trastuzumab
Period: Phase I - Core Phase
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Started | 6 | 17 | 10 | 0
Completed | 5 | 7 | 7 | 0
Not Completed | 1 | 10 | 3 | 0
Not completed — Disease Progression | 0 | 6 | 2 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: Phase I - Extension Phase
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Started | 5 | 7 | 7 | 0
Completed | 0 | 1 | 0 | 0
Not Completed | 5 | 6 | 7 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Disease Progression | 5 | 5 | 6 | 0
Period: Phase II - Core Phase
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Started | 0 | 0 | 0 | 55
Completed | 0 | 0 | 0 | 28
Not Completed | 0 | 0 | 0 | 27
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Disease Progression | 0 | 0 | 0 | 16
Not completed — Adverse Event | 0 | 0 | 0 | 8
Period: Phase II - Extension Phase
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Started | 0 | 0 | 0 | 24 (4 patients did not enter the Extension phase.)
Completed | 0 | 0 | 0 | 1 (Completed means 'Ongoing')
Not Completed | 0 | 0 | 0 | 23
Not completed — Disease Progression | 0 | 0 | 0 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all patients who received a least one dose of any one compound of the study treatment. Patients were analyzed according to the everolimus dose level to which they enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily | Total
Number analyzed (Participants) | 6 | 17 | 10 | 55 | 88
Age, Customized [Number; unit: Participants]
  Phase I : < 65 | 6 | 13 | 6 | 0 | 25
  Phase I : >= 65 | 0 | 4 | 4 | 0 | 8
  Phase II : < 65 | 0 | 0 | 0 | 49 | 49
  Phase II : >= 65 | 0 | 0 | 0 | 6 | 6
Sex/Gender, Customized [Number; unit: Participants]
  Phase I- Female | 6 | 17 | 10 | 0 | 33
  Phase II - Female | 0 | 0 | 0 | 55 | 55
Who Performance Status [Number; unit: Participants] — 0=Fully active, able to carry out normal activity without restriction, 1=Restricted in physical strenuous activity but ambulatory and able to carry work of a light or sedentary nature e.g. light house work, office work.
  Participants
    0 | 4 | 5 | 4 | 36 | 49
    1 | 2 | 12 | 6 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Overall Response Rate
Description: The primary objective of this phase II study was to evaluate the efficacy of the dose level/regimen of everolimus recommended from the Phase I with trastuzumab and paclitaxel (PT) therapy in patients with HER2-overexpressing metastatic breast cancer whose disease progressed on/after trastuzumab mono-and/or combination therapy based on the evaluation of objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Objective response rate (ORR) was defined as the proportion of patients with a best overall response (BOR) of complete response (CR) or partial response (PR). Only patients with measurable disease (the presence of at least one measurable lesion) at baseline were included in the study. CR = Disappearance of all target lesions; PR = At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: every 8 - 9 weeks until disease progression or a new lesion is identified
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Number analyzed (Participants) | 0 | 0 | 0 | 55
Percentage of Participants |  |  |  | 21.8

2. Secondary Outcome: Phase I: Best Overall Response (BOR)
Description: BOR was determined based on investigator assessment of overall lesion response using RECIST criteria guidelines. BOR = objective responses rate (ORR), disease control rate (DCR) or clinical benefit rate (CBR). ORR = (complete response (CR) or partial response(PR); DCR = (CR or PR or Stable disease (SD); CBR = (CR or PR or SD >= 24 weeks).CR = Disappearance of all target lesions; PR = At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for partial disease (PD). PD = At least a 20% increase in the sum of the longest diameter of all measured target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline.
Time Frame: every 8 - 9 weeks until disease progression or a new lesion is identified
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Number analyzed (Participants) | 6 | 17 | 10 | 0
Percentage of Participants
  Objective Response Rate (ORR) | 83.3 | 23.5 | 30.0 |
  Disease Control Rate (DCR) | 83.3 | 82.4 | 80.0 |
  Clinical Benefit Rate (CBR) | 83.3 | 47.1 | 70.0 |

3. Secondary Outcome: Phase II: Progression Free Survival (PFS)
Description: PFS is defined as the time from start of treatment to the date of first documented progression or death due to any cause. If a patient has not had an event, PFS will be censored at the date of last adequate tumor assessment.
Time Frame: every 8 - 9 weeks until disease progression or a new lesion is identified
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Number analyzed (Participants) | 0 | 0 | 0 | 55
Months |  |  |  | 5.52 [4.99 to 7.69]

4. Secondary Outcome: Phase II: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from start of treatment to the date of death due to any cause. If a patient is not known to have died, survival was censored at the last date of contact. OS was to be reported at extension and after 3-year follow-up. The Kaplan-Meier median was used to analyze the OS.
Time Frame: every 3 months until death
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I - RAD001 5mg + PT, Daily | Phase I - RAD001 10mg + PT, Daily | Phase I - RAD001 30mg + PT, Weekly | Phase II - RAD001 10mg + PT, Daily
Number analyzed (Participants) | 0 | 0 | 0 | 55
Months |  |  |  | 18.07 [12.85 to 24.11]

ADVERSE EVENTS:
Groups:
- Phase I - Everolimus 5mg Daily + PT; Phase I - Everolimus 10mg Daily + PT: Phase I - Daily dosing schedule of Everolimus 5mg plus Paclitaxel plus Trastuzumab. PT = Paclitaxel & Trastuzumab
- Phase I - Everolimus 30mg Weekly + PT: Phase I - Weekly dosing schedule of Everolimus 30mg plus Paclitaxel plus Trastuzumab. PT = Paclitaxel & Trastuzumab
- Phase II - Everolimus 10mg Daily + PT: Phase II - Daily dosing schedule of Everolimus 10mg plus Paclitaxel plus Trastuzumab. PT = Paclitaxel & Trastuzumab
Arm/Group | Phase I - Everolimus 5mg Daily + PT | Phase I - Everolimus 10mg Daily + PT | Phase I - Everolimus 30mg Weekly + PT | Phase II - Everolimus 10mg Daily + PT
Serious Adverse Events (participants affected / at risk) | 3/6 | 6/17 | 7/10 | 26/55
Other Adverse Events (participants affected / at risk) | 6/6 | 17/17 | 10/10 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Everolimus 5mg Daily + PT (N=6) | Phase I - Everolimus 10mg Daily + PT (N=17) | Phase I - Everolimus 30mg Weekly + PT (N=10) | Phase II - Everolimus 10mg Daily + PT (N=55)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Asthenia (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 6
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 2
Coma (Nervous system disorders) | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tracheal obstruction extrinsic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Everolimus 5mg Daily + PT (N=6) | Phase I - Everolimus 10mg Daily + PT (N=17) | Phase I - Everolimus 30mg Weekly + PT (N=10) | Phase II - Everolimus 10mg Daily + PT (N=55)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 4 | 19
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 9 | 2 | 12
Lymphopenia (Blood and lymphatic system disorders) | 2 | 7 | 5 | 11
Microcytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 12 | 5 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 9
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 3
Dry eye (Eye disorders) | 0 | 1 | 1 | 1
Eye inflammation (Eye disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 2 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 5
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 3 | 0 | 9
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 8 | 5 | 13
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 11 | 7 | 30
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 7 | 5 | 21
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 16 | 8 | 42
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 5 | 4 | 12
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 4 | 8 | 6 | 28
Chest pain (General disorders) | 0 | 1 | 1 | 2
Chills (General disorders) | 1 | 1 | 1 | 2
Face oedema (General disorders) | 0 | 0 | 0 | 3
Facial pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 3 | 12
Gait disturbance (General disorders) | 0 | 2 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 3
Oedema (General disorders) | 0 | 2 | 0 | 1
Oedema peripheral (General disorders) | 2 | 11 | 3 | 13
Pyrexia (General disorders) | 4 | 7 | 1 | 19
Xerosis (General disorders) | 0 | 2 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 2 | 0 | 1 | 2
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 1 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 3
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 2
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 2 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 2
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 4 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 2
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 4
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 10
Oral herpes (Infections and infestations) | 0 | 3 | 0 | 5
Oral infection (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 4
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 3 | 5 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 3 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 4
Urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 10
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 1
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 0 | 1 | 2
Echography abnormal (Investigations) | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 1 | 1 | 2
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 3 | 2 | 11
Weight increased (Investigations) | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 3 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 4
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 4
Dysaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 4
Headache (Nervous system disorders) | 1 | 8 | 3 | 23
Horner's syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 2
Hypokinesia (Nervous system disorders) | 0 | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 1 | 20
Neurotoxicity (Nervous system disorders) | 1 | 1 | 0 | 6
Paraesthesia (Nervous system disorders) | 2 | 6 | 4 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 1 | 3
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 4 | 2 | 6
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Genital discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2 | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 3 | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 6
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Tracheal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 6 | 5 | 15
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 10
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 6
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 6
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 5
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 8 | 3 | 26
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2
Lymphoedema (Vascular disorders) | 1 | 3 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.